CLINICAL TRIAL: NCT07222020
Title: Phase I, Placebo-Controlled, Double-Blinded, Randomized, Interventional, Safety and Pharmacokinetic Study of Single and Multiple Dosing of KB15A, a Vaginal Film Containing KB15A, an Anti-Sperm Monoclonal Antibody
Brief Title: Phase 1 Study of Intravaginal KB15A
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: ZabBio Inc. (Industry)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH); Boston University (Other); Old Dominion University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: KB15A-01; 5P50HD096957-08 (NIH)
Record Dates: First submitted 2025-10-24; First posted 2025-10-29 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Healthy Subjects

STUDY DESIGN:
Intervention Model Description: Placebo-Controlled, Double-Blinded, Randomized, Interventional
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- KB15A (Experimental): KB15A (Vaginal Film)
  Interventions: Drug: KB15A Vaginal Film
- Placebo (Placebo Comparator): Placebo (Vaginal Film)
  Interventions: Drug: Placebo Vaginal Film

INTERVENTIONS:
Drug: KB15A Vaginal Film — KB15A is a polyvinyl-alcohol based intravaginal film containing the KB15A.16.2 monoclonal antibody.
  Arms: KB15A
Drug: Placebo Vaginal Film — The Placebo is a polyvinyl-alcohol based intravaginal film composed identically to the KB15A Vaginal Film, but without the KB15A.16.2 monoclonal antibody.
  Arms: Placebo

SUMMARY:
The goal of this clinical trial is to determine the safety and mucosal pharmacokinetics of KB15A, a vaginal film containing an anti-sperm monoclonal antibody, in healthy adult women. Researchers will compare KB15A use to placebo use, primarily to see if KB15A is associated with adverse events, and also to understand the local and systemic distribution of the KB15A monoclonal antibody following use of the vaginal film.

Participants will be assessed for the genital, mucosal and systemic safety and pharmacokinetics of KB15A in a preliminary single-dose phase of the study, where they will receive two single doses of either KB15A or placebo vaginal film, and again in a multiple-dose phase of the study, where they will receive 14 daily doses of either KB15A or placebo vaginal film.

DETAILED DESCRIPTION:
KB15A is a polyvinyl-alcohol (PVA) based intravaginal contraceptive film Drug Product manufactured by KBio, Inc. containing the KB15A.16.2 Drug Substance. KB15A.16.2 is an IgG1 monoclonal antibody that targets CD52g, a unique glycan present on the surface of human sperm. KB15A is thought to work as a contraceptive by binding and trapping sperm in the vagina, so that they cannot migrate past the cervix and fertilize an oocyte.

This study will determine whether the KB15A film is safe in healthy women 18 - 45 years of age; it will also determine where the KB15A antibody is distributed in the body after film use. Participants must not be at risk of pregnancy due to one of the following approved methods of contraception or abstinence:

* prior surgical sterilization of self or sexual partner
* oral contraceptive pills
* transdermal patch
* contraceptive injection
* hormonal intrauterine system (IUS)
* heterosexual abstinence, or
* copper intrauterine device

Participants will be assessed for the genital, mucosal and systemic safety and pharmacokinetics of KB15A in two sequential study phases, separated by an approximately 2 - 6 week wash out period:

1. A preliminary single-dose phase of the study where participants will receive two single doses of either KB15A or placebo vaginal film, separated by approximately 1 week;
2. A multiple-dose phase of the study where participants will receive 14 consecutive daily doses of either KB15A or placebo vaginal film.

For the primary objective of the study, participants will be evaluated for Treatment Emergent Adverse Events (TEAEs) and relatedness of TEAEs to study product or study procedures, changes in colposcopic findings, and changes in systemic laboratories (e.g. complete blood count, chemistry panel) after two single doses in the single dose phase, and again after 14 daily doses in the multiple dose phase.

The secondary objective of the study is to describe the concentration of monoclonal antibody locally in the cervicovaginal mucosa, and systemically in the blood. Pharmacokinetics will be measured at baseline and at 30 minutes and 1, 2, and 4 hours after the first single dose; at 30 minutes and 8 or 48 hours after the second single dose (depending on the pharmacokinetic sampling time point randomization assignment); at 1, 4, 8, and 24 hours after the 1st dose of film in the multiple dose phase; and 24 hours after the 14th dose in the multiple dose phase. Finally, pharmacokinetics will be measured 5 - 8 days after the 14th dose of the film in the multiple-dose phase.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 to 45 years, inclusive
* General good health (by volunteer history and per investigator judgment) without any clinically significant systemic disease (including, but not limited to significant liver disease/hepatitis, gastrointestinal disease, kidney disease, thyroid disease, osteoporosis or bone disease, and diabetes) and with an intact gastrointestinal tract, uterus and cervix.
* History of regular menstrual cycles, by volunteer report, if not taking exogenous hormones
* History of Pap smears and follow-up consistent with standard clinical practice as outlined in the Study Manual or willing to undergo a Pap smear at Visit 1
* Willing to give voluntary consent and sign an informed consent form.
* Willing to use non-spermicidal, lubricated condoms for any vaginal intercourse according to the study protocol.
* Willing to abstain from intercourse and use of intravaginal medications, lubricants, and other products as required in the protocol.
* Vaginal and cervical anatomy that, in the opinion of the investigator, lends itself to easy genital tract sample collection.
* Must be protected from pregnancy by:

  * Sterilization of either partner
  * Heterosexual abstinence
  * Hormonal contraceptives (except for the contraceptive vaginal ring)
  * Copper IUD
* If in a relationship, must be in a mutually monogamous relationship with a partner who is not known to be HIV positive and has no known risk of sexually transmitted infections (STIs)

Exclusion Criteria:

* History of hysterectomy
* Currently pregnant
* Currently breastfeeding or planning to breastfeed during the course of the study
* Current Positive test for Trichomonas vaginalis, Neisseria gonorrhea, Chlamydia trachomatis,
* Current symptomatic bacterial vaginosis (BV)
* Chronic or acute vulvar or vaginal symptoms (pain, irritation, spotting/bleeding, discharge, etc.)
* Significant gynecological abnormalities (including abnormal vaginal bleeding, excessive vaginal discharge, or vulvar/vaginal pain or irritation)
* Current symptomatic UTI or vaginal candidiasis
* History of sensitivity/allergy to KB15A film components, for either the volunteer
* Less than 14 days since use of oral or vaginal antibiotics
* Women with a history of genital herpes or condylomata who have been symptomatic in the last six months.
* Deep epithelial genital findings such as abrasions, ulcerations, and lacerations, or vesicles suspicious for an STI
* Known current drug or alcohol abuse which could affect study compliance.
* Participation in any other investigational trial within the last 30 days or planned participation in any other investigational trial during the study
* History of gynecological procedures (including genital piercing) on the external genitalia, vagina or cervix within the last 14 days
* Abnormal finding on laboratory or physical examination or a social or medical condition in the participant, which, in the opinion of the investigator, would make participation in the study unsafe or would complicate interpretation of data.
* Grade 2 or higher laboratory abnormality, per the 2014 update of the Division of AIDS, National Institute of Allergy and Infectious Disease (DAIDS) Table for Grading the Severity of Adverse Events, or clinically significant laboratory abnormality as determined by the clinician.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2026-09-01 (Estimated); Study Completion 2026-12-28 (Estimated)

PRIMARY OUTCOMES:
Treatment Emergent Adverse Events (TEAEs) and relatedness of TEAEs to study product or study procedures. | From baseline through study completion, on average 3-4 months
Change in colposcopic findings | From baseline through study completion, on average 3-4 months
Number of Participants With Abnormal Laboratory Values | From baseline through study completion, on average 3-4 months

SECONDARY OUTCOMES:
Mass of anti-sperm-antibody in the vagina | Baseline; 30 minutes, 1, 2 and, 4 hours after first single dose; 30 minutes and 8 or 48 hours after second single dose; 1, 4, 8 and 24 hours after first multi-dose; and 24 hours and 5 - 8 days after final multi-dose.
  Mass of anti-sperm-antibody in the cervicovaginal fluid from vaginal swabs and cervicovaginal fluid lavage (CVL) supernatant.
Concentration of anti-sperm-antibody in serum | Baseline; 48 hours after first single dose; 48 hours after second single dose; and 24 hours after final multi-dose

CONTACTS AND LOCATIONS:
Locations (1):
- Virginia Health Sciences at Old Dominion University, Norfolk, Virginia, United States

IPD SHARING:
Plan to Share IPD: No